CLINICAL TRIAL: NCT01286402
Title: Double-blind, Placebo-Controlled Pilot Study of Bupropion to Promote Smoking Cessation During Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Gilstrap, Larry C, M.D. (Individual); The Center for Clinical and Translational Sciences (CCTS) Clinical Research Unit at The University of Texas Health Science Center at Houston (Other)
Responsible Party: Principal Investigator, Angela Stotts, Associate Professor - Family Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-09-0681
Record Dates: First submitted 2011-01-25; First posted 2011-01-31 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation during pregnancy; bupropion
MeSH Terms: conditions — Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion SR (sustained release) (Experimental): Group receiving bupropion SR medication
  Interventions: Drug: Bupropion SR
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupropion SR — * 150mg, taken orally, taken daily for the 1st 3 days
  * 300mg, taken orally, taken daily for the rest of the 8 weeks of drug treatment
  Other Names: Zyban, Wellbutrin
  Arms: Bupropion SR (sustained release)
Other: Placebo — -Avicel PH 302, Emcocel 50M, Cab-O-Sil M5P, Magnesium Stearate (appearance, taste, and dosing instructions were identical to the bupropion group), i.e., 1 pill orally, taken daily for the 1st 3 days; 2 pills, taken orally, taken daily for the rest of the 8 weeks of drug treatment
  Arms: Placebo

SUMMARY:
This study is designed to gather preliminary effectiveness and safety data on the use of bupropion for smoking cessation in pregnant women attending a community prenatal clinic. This study will provide critical preliminary data in preparation for a larger, Phase III clinical trial.

DETAILED DESCRIPTION:
A randomized, double-blind, parallel group design will be used to allow a rigorous preliminary assessment of the feasibility, effectiveness, and safety of bupropion SR (sustained release; packaged as Zyban by GlaxoSmithKline) in promoting smoking cessation among women in their second and third trimester of pregnancy. Fifty pregnant smokers will be randomized to receive an 8-week course of either bupropion SR or matching placebo tablets. Both groups will receive evidence-based smoking cessation counseling. The primary smoking outcome will be 7-day point prevalence abstinence with cotinine validation at the end of the treatment. Secondary outcomes include enrollment, retention, and compliance rates; continuous abstinence from end of treatment through the 2 week followup; continuous abstinence from birth to 2nd week postpartum followup; self-reported reduction in number of cigarettes smoked per day; and maternal side effects and perinatal/neonatal outcomes. Preliminary smoking cessation and safety outcomes will be assessed for the generation of evidence-based hypotheses regarding clinical benefit of bupropion for pregnant smokers in preparation fo a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 18 years of age
* Gestational age between 14 and 26 weeks confirmed by ultrasound
* Currently smoking ≥ 5 cigarettes per day

Exclusion Criteria:

* Abnormal liver function tests
* History of or current seizure disorder or closed head injury with loss of consciousness
* Known hypersensitivity to bupropion
* Any psychiatric disorder requiring psychotropic medication
* Current anorexia or bulimia
* Use of monoamine oxidase (MAO) inhibitors or discontinuation within the past 2 weeks
* Major Depressive Disorder or current suicidal risk
* Use of any illicit substances since receiving knowledge of pregnancy
* Regular use of alcohol (>1 drink/week on average)
* Unstable medical problems, such as liver or renal disease, uncontrollable hypertension, and lupus
* Twins or other multiple gestation
* Fetal abnormality on the 14 week ultrasound
* Plans to deliver at a hospital other than Memorial Hermann
* Inability to communicate with research staff or make study visits due to lack of phone or transportation access
* Participation in another clinical study which may affect study outcomes
* Current use of any Nicotine Replacement Therapy (NRT), bupropion, or varenicline (Chantix)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Stotts, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Professional Building, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion SR (Sustained Release): Group receiving bupropion SR medication
  Bupropion SR: - 150mg (1 pill), taken orally, taken daily for the 1st 3 days
  - 300mg (2 pills), taken orally, taken daily for the rest of the 8 weeks of drug treatment
- Placebo: Group receiving placebo
  -Avicel PH 302, Emcocel 50M, Cab-O-Sil M5P, Magnesium Stearate (appearance, taste, and dosing instructions were identical to the bupropion group), i.e., 1 pill orally, taken daily for the 1st 3 days; 2 pills, taken orally, taken daily for the rest of the 8 weeks of drug treatment
Period: Overall Study
Arm/Group | Bupropion SR (Sustained Release) | Placebo
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bupropion SR (Sustained Release): Group receiving bupropion SR medication
  Bupropion SR: - 150mg, taken orally, taken daily for the 1st 3 days
  - 300mg, taken orally, taken daily for the rest of the 8 weeks of drug treatment
- Total: Total of all reporting groups
Arm/Group | Bupropion SR (Sustained Release) | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (5.6) | 26.7 (5.9) | 26.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
# cigs smoked in past 30 days [Mean (Standard Deviation); unit: cigarettes] | 10.8 (11.1) | 10.7 (5.4) | 10.7 (8.0)
Age started smoking [Mean (Standard Deviation); unit: years] | 17.8 (3.0) | 17.3 (9.0) | 17.5 (4.3)
Carbon monoxide reading [Mean (Standard Deviation); unit: parts per million] | 8.8 (3.7) | 15.2 (17.5) | 12.0 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Smoking Abstinence With Cotinine Validation at the End of Treatment
Time Frame: 1 week post treatment
Measure: Number; unit: participants
Arm/Group | Bupropion SR (Sustained Release) | Placebo
Number analyzed (Participants) | 5 | 6
participants | 0 | 2

2. Secondary Outcome: Enrollment, Retention and Compliance Rates
Time Frame: 1 year (estimated)
Reporting Status: Not Posted

3. Secondary Outcome: Continuous Abstinence From End of Treatment Through the 2 Week Followup
Time Frame: at two week followup visit
Reporting Status: Not Posted

4. Secondary Outcome: Continuous Abstinence From Birth to 2nd Week Postpartum Followup
Time Frame: at 2nd week postpartum followup visit
Reporting Status: Not Posted

5. Secondary Outcome: Self-reported Reduction in Number of Cigarettes Smoked Per Day
Time Frame: at 1 week post treatment and at 2 week postpartum visit
Reporting Status: Not Posted

6. Secondary Outcome: Maternal Side Effects
Time Frame: during treatment, end of treatment and at 2 week postpartum visit
Reporting Status: Not Posted

7. Secondary Outcome: Perinatal/Neonatal Outcomes
Time Frame: at neonatal discharge from hospital following delivery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bupropion SR (Sustained Release) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/6
Other Adverse Events (participants affected / at risk) | 2/5 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion SR (Sustained Release) (N=5) | Placebo (N=6)
Newborn readmission for respiratory failure on day of life 5 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — MOTHER HAD UPPER RESPIRATORY SYMPTOMS SUGGESTIVE OF INFECTION. INFANT HAD DECREASED FEEDING, LETHARY, DEHYDRATION AND DEVELOPED APNOEA AND WAS INTUBATED FOR RESPIRATORY SUPPORT. EVENT THOUGHT NOT BE RELATED TO STUDY MEDICATION AND IS RESOLVED.
Hyperbilirubinemia secondary to ABO incompatibility (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion SR (Sustained Release) (N=5) | Placebo (N=6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No